CLINICAL TRIAL: NCT02595398
Title: A Phase 3, Randomized, Masked, Controlled Clinical Trial to Study the Safety and Efficacy of Triamcinolone Acetonide Injectable Suspension (CLS-TA) for the Treatment of Subjects With Macular Edema Associated With Non-infectious Uveitis
Brief Title: Suprachoroidal Injection of CLS-TA in Subjects With Macular Edema Associated With Non-infectious Uveitis
Acronym: PEACHTREE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS1001-301
Record Dates: First submitted 2015-10-28; First posted 2015-11-03 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Uveitis; Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate; Panuveitis
Keywords: Uveitis; UME; Posterior Uveitis; Anterior Uveitis; Intermediate Uveitis; Panuveitis; Non-infectious Uveitis; Triamcinolone; Choroid; Choroidal Injection; Suprachoroidal; Microneedle; Microinjection; Triamcinolone acetonide
MeSH Terms: conditions — Uveitis; Uveitis, Posterior; Uveitis, Anterior; Uveitis, Intermediate; Panuveitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4mg CLS-TA Suprachoriodal Injection (Experimental): Suprachoroidal injection of 40 mg/mL (4 mg in 100 µL) of CLS-TA
  Interventions: Drug: 4mg CLS-TA Suprachoriodal Injection
- Sham Procedure (Sham Comparator): Matching suprachoroidal syringe with sham procedure
  Interventions: Drug: Sham Procedure

INTERVENTIONS:
Drug: 4mg CLS-TA Suprachoriodal Injection — CLS-TA, 40 mg/mL (4 mg in 100 µL), administered as a single injection at 2 timepoints
  Other Names: Triamcinolone Acetonide
  Arms: 4mg CLS-TA Suprachoriodal Injection
Drug: Sham Procedure — Sham procedure administered at 2 timepoints
  Other Names: suprachoroidal sham
  Arms: Sham Procedure

SUMMARY:
The study is designed to evaluate the safety and efficacy of suprachoroidally administered triamcinolone acetonide, CLS-TA, in subjects with macular edema associated with non-infectious uveitis.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, masked, sham-controlled, multicenter study to assess the safety and efficacy of 4 mg of CLS-TA administered via suprachoroidal injection compared to a sham injection procedure in the treatment of subjects with macular edema associated with non-infectious uveitis.

Qualified subjects will be randomized to receive two suprachoroidal injections of CLS-TA administered to the study eye or two sham injection procedures administered to the study eye approximately 12 weeks apart (Visit 2 and Visit 5). Follow-up visits will be conducted monthly up to 24 weeks (Visit 8).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-infectious uveitis (pan, anterior, intermediate and posterior)
* Diagnosis of macular edema associated with non-infectious uveitis (retinal thickness ≥ 300 microns)
* Visual Acuity score of ≥ 5 letters read (20/800 Snellen equivalent) and ≤ 70 letters read (20/40 Snellen equivalent), in the study eye

Exclusion Criteria:

* Any active ocular disease or infection in the study eye other than uveitis
* Intraocular pressure > 22 mmHg or uncontrolled glaucoma in the study eye; subjects are not excluded if IOP ≤ 22 mmHg with no more than 2 IOP lowering medications.
* Any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study
* Any topical ocular corticosteroid in the 10 days prior to baseline; intraocular or periocular corticosteroid injections in the 2 months prior to baseline; an OZURDEX implant in the 6 months prior to baseline; RETISERT or ILUVIEN implant in the 3 years prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cuilla, MD, MBA, Study Director — Clearside Biomedical, Inc.
Locations (64):
- United States (40):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina Centers, PC, Tucson, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - USC Eye Institute, Los Angeles, California
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - Orange County Retina Medical Group, Santa Ana, California
  - University of Colorado, Aurora, Colorado
  - Colorado Retina Associates, Golden, Colorado
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Center for Retina and Macular Disease, Lakeland, Florida
  - Emory Eye Center Emory University, Atlanta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Illinois Retina Associates, S.C., Oak Park, Illinois
  - Midwest Eye Retina Practicing at Midwest Eye Institute, Indianapolis, Indiana
  - Elman Retina Group, PA, Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Valley Eye Physicians and Surgeons, PC, Ayer, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Ocular Immunology and Uveitis Foundation; Massachusetts Eye Research and Surgery Institution, Waltham, Massachusetts
  - Discover Vision Centers, Independence, Missouri
  - Metropolitan Eye Research & Surgery Institute, Palisades Park, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Retina Consultants PLLC, Slingerlands, New York
  - Charlotte Eye Ear Nose and Throat Associates, PA, Belmont, North Carolina
  - Wake Forest Baptist Health Eye Center, Winston-Salem, North Carolina
  - Bergstrom Eye Research, Fargo, North Dakota
  - Oregon Health & Science University Casey Eye Institute, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Eye Center, Pittsburgh, Pennsylvania
  - Innovative Clinical Research, Greenville, South Carolina
  - Austin Retina Associates, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Foresight Studies, LLC, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
  - Vitreoretinal Associates of Washington, Bellevue, Washington
- India (16):
  - L V Prasad Eye Hospital, Hyderabad, Andhra Pradesh
  - Sri Sankaradeva Nethralaya, Guwahati, Assam
  - M&J Western Regional Institute of Ophthalmology, Ahmedabad, Gujarat
  - JSS Hospital, Mysore, Karnataka
  - Regional Institute of Ophthalmology, Thiruvananthapuram, Kerala
  - TN Medical College and BYL Nair Hospital, Mumbai, Maharashtra
  - PBMA's H V Desai Eye Hospital, Pune, Maharashtra
  - Sankara Nethralaya, Chennai, Tamil Nadu
  - Sankara Eye Hospital, Coimbatore, Tamil Nadu
  - King George's Medical University, Lucknow, Uttar Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Icare Eye Hospital & PG Institute, Noida, Uttar Pradesh
  - Calcutta Medical Research Institute, Kolkata
  - Disha Eye Hospital, Kolkata
  - Dr Rajendra Prasad Centre for Ophthalmic Sciences, New Delhi
  - Dr. Shroff's Charity Eye Hospital, New Delhi
- Israel (8):
  - Soroka Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Corp, Haifa
  - Hadassah-Hebrew University Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeh S, Ciulla T. Suprachoroidal triamcinolone acetonide injectable suspension for macular edema associated with noninfectious uveitis: an in-depth look at efficacy and safety. Am J Manag Care. 2023 Feb;29(2 Suppl):S19-S28. doi: 10.37765/ajmc.2023.89324. PMID 36787524
- [Derived] Yeh S, Henry CR, Kapik B, Ciulla TA. Triamcinolone Acetonide Suprachoroidal Injectable Suspension for Uveitic Macular Edema: Integrated Analysis of Two Phase 3 Studies. Ophthalmol Ther. 2023 Feb;12(1):577-591. doi: 10.1007/s40123-022-00603-x. Epub 2022 Nov 18. PMID 36399237
- [Derived] Bhattacharyya S, Hariprasad SM, Albini TA, Dutta SK, John D, Padula WV, Harrison D, Joseph G. Suprachoroidal Injection of Triamcinolone Acetonide Injectable Suspension for the Treatment of Macular Edema Associated With Uveitis in the United States: A Cost-Effectiveness Analysis. Value Health. 2022 Oct;25(10):1705-1716. doi: 10.1016/j.jval.2022.07.008. Epub 2022 Aug 31. PMID 36055922
- [Derived] Singer MA, Merrill P, Yeh S, Hall C, Kapik B, Ciulla TA. Suprachoroidal triamcinolone acetonide versus rescue therapies for the treatment of uveitic macular oedema: A post hoc analysis of PEACHTREE. Clin Exp Ophthalmol. 2022 Jan;50(1):23-30. doi: 10.1111/ceo.14024. Epub 2021 Dec 27. PMID 34741564
- [Derived] Price KW, Albini TA, Yeh S. Suprachoroidal Injection of Triamcinolone- Review of a Novel Treatment for Macular Edema Caused by Noninfectious Uveitis. US Ophthalmic Rev. 2020 Fall;13(2):76-79. doi: 10.17925/usor.2020.13.2.76. Epub 2020 Dec 23. PMID 34322164

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4mg CLS-TA Suprachoriodal Injection | Sham Procedure
Started | 96 | 64
Intention-to-Treat (ITT) Population (Defined as all randomized subjects who received at least one study treatment. Subjects analyzed as originally allocated after randomization.) | 96 | 64
Safety Population (Defined as all randomized subjects who were administered at least one dose of study drug.) | 96 | 64
Completed | 92 | 63
Not Completed | 4 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat population included all randomized subjects who received at least one study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 4mg CLS-TA Suprachoriodal Injection | Sham Procedure | Total
Number analyzed (Participants) | 96 | 64 | 160
Age, Categorical [Count of Participants; unit: Participants] — Age of subjects in years relative to the date of the Screening visit.
  Participants
    <=18 years | 1 | 0 | 1
    Between 18 and 65 years | 79 | 52 | 131
    >=65 years | 16 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of subjects in years relative to the date of the Screening visit.
  years | 50.40 (14.180) | 50.00 (15.083) | 50.24 (14.502)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 34 | 88
  Male | 42 | 30 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 86 | 58 | 144
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 44 | 28 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 40 | 25 | 65
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 34 | 80
  Israel | 7 | 3 | 10
  India | 43 | 27 | 70
Type of Uveitis [Count of Participants; unit: Participants] — Location of inflammation in the study eye, including anterior (anterior chamber), intermediate (vitreous), posterior (retina or choroid) and panuveitis.
  Participants
    Anterior uveitis | 27 | 14 | 41
    Intermediate uveitis | 34 | 23 | 57
    Posterior uveitis | 22 | 13 | 35
    Panuveitis | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Demonstrating ≥ 15 Letter Improvement From Baseline in Best Corrected Visual Acuity at 24 Weeks
Description: Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured in the number of letters read correctly on electronic Visual Acuity (eVA). An increase from the pre-treatment state in BCVA of 15 letters or more represents a clinically meaningful improvement.
Time Frame: Baseline, 24 weeks
Population: The Intent-to-treat population included all randomized subjects who received at least one study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 4mg CLS-TA Suprachoriodal Injection | Sham Procedure
Number analyzed (Participants) | 96 | 64
Participants | 45 | 10
Statistical Analysis 1: Comparison: 4mg CLS-TA Suprachoriodal Injection vs Sham Procedure; A total sample size of 150 subjects in a 3:2 randomization had 90% power to detect a difference between treatments in the proportion of subjects showing improvement is 0.60 for treated and 0.34 for sham. The primary analysis was a test of superiority of the CLS-TA arm over the sham arm, and was based on a Cochran-Mantel-Haenszel chi-square test stratified by country; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The a priori threshold for statistical significance was 0.050. Prior to evaluating the results of the CMH test, a Breslow-Day test with Tarone's adjustment was conducted to confirm the homogeneity of the odds ratios between country strata; The CMH test was stratified by the country, i.e., US+Israel and India; Difference in percentages = 31.25, 95% CI 2-sided [15.5 to 45.9] — Estimated value was calculated as the percentage of subjects in the Active arm meeting the primary endpoint minus the percentage of subjects in the Control arm meeting the primary endpoint

2. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness
Description: Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A masked reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema. Only images that were gradable by the central reading center were included in the analysis.
Time Frame: Baseline, 24 weeks
Population: The Intent-to-treat population included all randomized subjects who received at least one study treatment. Analysis included all subjects with gradable reading center images.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | 4mg CLS-TA Suprachoriodal Injection | Sham Procedure
Number analyzed (Participants) | 93 | 61
microns | -152.6 (159.14) | -17.9 (150.98)

3. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Number of subjects with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) reported between the first dose of study drug and study exit.
Time Frame: Baseline to 24 weeks
Population: The Safety population included all randomized subjects who were administered at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 4mg CLS-TA Suprachoriodal Injection | Sham Procedure
Number analyzed (Participants) | 96 | 64
Participants
  Experiencing at least one TEAE | 67 | 45
  Experiencing at least one SAE | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 24 weeks of follow-up.
Arm/Group | 4mg CLS-TA Suprachoriodal Injection | Sham Procedure
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/64
Serious Adverse Events (participants affected / at risk) | 3/96 | 0/64
Other Adverse Events (participants affected / at risk) | 42/96 | 29/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4mg CLS-TA Suprachoriodal Injection (N=96) | Sham Procedure (N=64)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4mg CLS-TA Suprachoriodal Injection (N=96) | Sham Procedure (N=64)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Cataract subcapsular (Eye disorders) | 7 (7) | 3 (4) — #Study eye
Cystoid macular oedema (Eye disorders) | 0 (0) | 9 (11) — #Study eye
Eye pain (Eye disorders) | 14 (18) | 0 (0) — #Study eye
Ocular hypertension (Eye disorders) | 2 (3) | 5 (5) — #Study eye
Uveitis (Eye disorders) | 2 (2) | 4 (4) — #Study eye
Intraocular pressure increased (Investigations) | 17 (21) | 4 (4) — #Study eye
Intraocular pressure increased (Investigations) | 6 (6) | 2 (2) — #Fellow eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02595398/Prot_SAP_000.pdf